CLINICAL TRIAL: NCT05937022
Title: Utilizing Transcranial Direct Current Stimulation (tDCS) to Boost Social Pleasure and Participation in Older Lonely Individuals
Brief Title: The Effects of Transcranial Direct Current Stimulation (tDCS) in Older Lonely Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Tatia Mei-chun LEE, Director, State Key Laboratory of Brain and Cognitive Sciences; Chair Professor of Psychological Science and Clinical Psychology; May Endowed Professor in Neuropsychology., The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: hkutdcsage
Record Dates: First submitted 2023-06-08; First posted 2023-07-10 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Loneliness
Keywords: Transcranial Direct Current Stimulation; Emotion Regulation; Lateral Prefrontal Cortex; Aging
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Participants are assigned to three groups in parallel for the duration of the study.
Who Masked: Participant
Masking Description: Participants will be unaware of their group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Right VLPFC tDCS (Experimental): Participants who are assigned to the right VLPFC group will receive anodal tDCS over the right ventrolateral prefrontal cortex (VLPFC).
  Interventions: Device: Experimental Transcranial Direct Current Stimulation (tDCS)
- Left DLPFC tDCS (Experimental): Participants who are assigned to the right VLPFC group will receive anodal tDCS over the left dorsolateral prefrontal cortex (DLPFC).
  Interventions: Device: Experimental Transcranial Direct Current Stimulation (tDCS)
- Sham Control tDCS (Sham Comparator): For the sham protocol, the electrode positioning will be randomly allocated to be identical to either the left DLPFC or the right VLPFC group, but the active stimulation will be delivered for the first 30 seconds only.
  Interventions: Device: Sham Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Experimental Transcranial Direct Current Stimulation (tDCS) — This study will deliver tDCS sessions for ten sessions completed within two weeks. Consecutive tDCS sessions are separated by at least 24 hours. Participants assigned to one of the two experimental groups will receive 20 minutes of active stimulation with a 2mA intensity over the corresponding brain regions.
  Arms: Left DLPFC tDCS; Right VLPFC tDCS
Device: Sham Transcranial Direct Current Stimulation (tDCS) — This study will deliver tDCS sessions for ten sessions completed within two weeks. Consecutive tDCS sessions are separated by at least 24 hours. Participants assigned to the sham control group will receive 30 seconds of active stimulation over brain regions identical to either the left DLPFC or the right VLPFC experimental tDCS group.
  Arms: Sham Control tDCS

SUMMARY:
This randomized clinical trial aims to test the effects of 10 sessions of transcranial direct current stimulation (tDCS) on social and emotional functions in lonely older adults.

The main objectives include:

* Understand whether tDCS could successfully boost positive social processing and social motivation in older adults, paralleling its effect on non-social reward processing;
* Understand whether the reduced negative and increased positive social processing in older adults would translate to an increase in real-life social activity and a decrease in loneliness feeling;
* Examine the intervention efficacy of tDCS among the aged population;
* Understand whether the tDCS effect could be long-lasting (i.e., 1 and 3 months after intervention).

Participants will be lonely older adults aged 60 or above and screened on inclusion and exclusion criteria. Eligible participants will be randomly allocated to the left dorsolateral prefrontal cortex (DLPFC) tDCS group, the right ventrolateral prefrontal cortex (VLPFC) tDCS group, or the sham control group. Participants will complete an Emotion Rating Task, questionnaires assessing their psychosocial functions, and neuropsychological tests assessing their cognitive functions at baseline, after the 5th stimulation session, immediately after the 10th stimulation session, and 1 month and 3 months after the 10th stimulation session.

DETAILED DESCRIPTION:
Loneliness, or perceived social isolation, results from discrepancies between an individual's desired and achieved social needs. A substantial proportion of older adults experience loneliness. With the social distancing policies implemented during the COVID-19 pandemic, older adults, who are more likely to be functionally dependent on their caregivers, have been primarily affected, contributing to adverse impacts on their social and emotional functions. As current loneliness interventions have shown limited efficacy, it is of great significance to test novel interventions for lonely older adults.

Transcranial direct current stimulation (tDCS) is a neuromodulatory technique that has demonstrated its safety and efficacy in modulating cortical excitability and associated behaviors in older adults. It has been suggested that repeated tDCS sessions show sustained therapeutic efficacy in chronic disorders. Additionally, the efficacy of tDCS as an intervention for lonely older adults has not been investigated. As a result, it is crucial to test repeated tDCS sessions as a potential intervention to reduce loneliness and improve socioemotional functions in lonely older adults.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 60 years old;
2. Fluent in reading and speaking Traditional Chinese (Cantonese or Mandarin);
3. Right-handed as assessed with the Edinburgh Handedness Inventory;
4. Normal or corrected-to-normal vision and hearing;
5. Normal general cognitive function as determined by the Hong Kong version of the Montreal Cognitive Assessment (HK-MoCA) ≥ 22;
6. ≥ 9 years of formal education as lexical comprehension is required in the Emotion Rating Task.

Exclusion Criteria:

1. Current or past major physical or neurological illness that significantly affects the individual's current cognitive, motor, or brain function;
2. Medication or other treatment received within 2 weeks before the study that may affect the individual's current cognitive, motor, or brain function;
3. Receiving maintained therapy that may affect cognitive, motor, or brain function and cannot be discontinued for the entire course of study;
4. Past or present major psychological conditions, including affective disorders, anxiety disorder, psychotic disorder, addiction, and impulse control disorder;
5. Any contraindication of tDCS, such as a cerebral implant or history (either personal or family) of seizure.
6. Participation in similar brain stimulation studies within the past six months.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2022-12-03 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in emotion and social motivation in response to social and non-social emotional stimuli | From baseline to after the 5th tDCS session (1 week); from baseline to after the 10th tDCS session (2 weeks); from baseline to 1 month after the last tDCS session; from baseline to 3 months after the last tDCS session.
  The Emotion Rating Task will assess participants' feelings and motivations upon seeing positive, negative, social, and non-social emotional words. Participants will need to rate on a scale regarding his/her emotional feelings and socializing motivation upon perceiving these words.
Changes in self-reported loneliness levels | From baseline to after the 5th tDCS session (1 week); from baseline to after the 10th tDCS session (2 weeks); from baseline to 1 month after the last tDCS session; from baseline to 3 months after the last tDCS session.
  Perceived level of loneliness will be assessed with the brief 6-item UCLA Loneliness Scale. All items are scored on a 4-point scale ranging from 1 (never) to 4 (often). The total score ranges from 6 to 24. A higher score indicates a higher level of perceived loneliness.

SECONDARY OUTCOMES:
Changes in social motivation | From baseline to after the 5th tDCS session (1 week); from baseline to after the 10th tDCS session (2 weeks); from baseline to 1 month after the last tDCS session; from baseline to 3 months after the last tDCS session.
  Participants' information-seeking and emotion-regulatory motivation will be measured with the Social Motivation Questionnaire (SMQ).
Changes in social anhedonia | From baseline to after the 5th tDCS session (1 week); from baseline to after the 10th tDCS session (2 weeks); from baseline to 1 month after the last tDCS session; from baseline to 3 months after the last tDCS session.
  The Dimensional Anhedonia Rating Scale (DARS) will assess participants' anhedonia in aspects including hobbies, dood/drink, social activities, and sensory experience. The participants will be instructed to provide at least two of their own examples for each pleasure domain. Participants will then be asked to rate items from 0 to 4 on a scale of not at all, slightly, moderately, mostly, and very much for each domain, with a lower score corresponding to a higher level of anhedonia.
Changes in social participation | From baseline to after the 10th tDCS session (2 weeks); from baseline to 1 month after the last tDCS session; from baseline to 3 months after the last tDCS session.
  The Participation Measure--3 Domains, 4 Dimensions (PM-3D4D) will assess participants' social participation.
Changes in perceived social support | From baseline to after the 5th tDCS session (1 week); from baseline to after the 10th tDCS session (2 weeks); from baseline to 1 month after the last tDCS session; from baseline to 3 months after the last tDCS session.
  The Multidimensional Scale of Perceived Social Support (MSPSS) will assess participants' perceived social support. This scale includes 3 subscales: significant other, family, and friends. The mean score of the total scale can be obtained by summing across all 12 items and then dividing by 12. A higher score on the scale means a higher level of perceived social support.
Changes in social isolation | From baseline to after the 10th tDCS session (2 weeks); from baseline to 1 month after the last tDCS session; from baseline to 3 months after the last tDCS session.
  The Abbreviated Lubben Social Network Scale (LSNS-6) will assess participants' social network size. The total score is the sum of the 6 items. Scores range from 0 to 30. A higher score indicates a lower level of social isolation.
Changes in positive and negative affect | From baseline to after the 5th tDCS session (1 week); from baseline to after the 10th tDCS session (2 weeks); from baseline to 1 month after the last tDCS session; from baseline to 3 months after the last tDCS session.
  Participants' emotional disposition and mood state will be measured with the Chinese Affect Scale (CAS). Participants will be instructed to rate on a scale from 0 to 4, with a higher score corresponding to a higher level of positive or negative affect. Scores of positive affect range from 0 to 40. Scores of negative affect range from 0 to 40.
Changes in emotion regulation | From baseline to after the 5th tDCS session (1 week); from baseline to after the 10th tDCS session (2 weeks); from baseline to 1 month after the last tDCS session; from baseline to 3 months after the last tDCS session.
  The Cognitive Emotion Regulation Questionnaire (CERQ) will assess participants' use of nine cognitive emotion regulation strategies.
Changes in coping styles | From baseline to after the 5th tDCS session (1 week); from baseline to after the 10th tDCS session (2 weeks); from baseline to 1 month after the last tDCS session; from baseline to 3 months after the last tDCS session.
  Coping Orientation to Problems Experienced Inventory (Brief-COPE) will assess participants' coping styles.
Changes in approach and avoidance motivation | From baseline to after the 5th tDCS session (1 week); from baseline to after the 10th tDCS session (2 weeks); from baseline to 1 month after the last tDCS session; from baseline to 3 months after the last tDCS session.
  Participants' reward responsiveness, drive, fun-seeking, and punishment sensitivity will be assessed with the behavioral inhibition system and behavioral activation system (BIS/BAS) scale. The scale consists of 18 items that are rated on a 4-point Likert scale, with 1 = strongly disagree, 2 = disagree, 3 = agree, and 4 = strongly agree. Scores are calculated as the sum of respective items. A higher score indicates a higher approach or avoidance motivation.
Changes in levels of depression | From baseline to after the 5th tDCS session (1 week); from baseline to after the 10th tDCS session (2 weeks); from baseline to 1 month after the last tDCS session; from baseline to 3 months after the last tDCS session.
  The Geriatric Depression Scale (GDS) will assess participants' levels of depression. Scores range from 0 to 30, with a higher score indicating a higher level of depression.
Changes in levels of anxiety | From baseline to after the 5th tDCS session (1 week); from baseline to after the 10th tDCS session (2 weeks); from baseline to 1 month after the last tDCS session; from baseline to 3 months after the last tDCS session.
  The Geriatric Anxiety Scale - 10 Item Version (GAS-10) will assess participants' anxiety levels. Items 1 through 10 are summed to provide a total score. Each item ranges from 0 to 3. The total score ranges from 0 to 30.
Changes in cognitive control functions | From baseline to after the 5th tDCS session (1 week); from baseline to after the 10th tDCS session (2 weeks); from baseline to 1 month after the last tDCS session; from baseline to 3 months after the last tDCS session.
  Cognitive control functions, specifically selective attention, will be assessed with the Chinese version (CST) of the Stroop Color Word Test (Victoria version).
Changes in processing speed | From baseline to after the 5th tDCS session (1 week); from baseline to after the 10th tDCS session (2 weeks); from baseline to 1 month after the last tDCS session; from baseline to 3 months after the last tDCS session.
  Processing Speed will be assessed with the Symbol Digit Modalities Test (SDMT).
Changes in working memory | From baseline to after the 5th tDCS session (1 week); from baseline to after the 10th tDCS session (2 weeks); from baseline to 1 month after the last tDCS session; from baseline to 3 months after the last tDCS session.
  The Digit Span Backward Test will assess working memory.
Changes in perceived levels of social and emotional loneliness | From baseline to after the 5th tDCS session (1 week); from baseline to after the 10th tDCS session (2 weeks); from baseline to 1 month after the last tDCS session; from baseline to 3 months after the last tDCS session.
  The self-reported social and emotional loneliness levels will be measured with the 6-item De Jong Gierveld Loneliness Scale. On the negatively worded items (1 to 3, emotional loneliness), the neutral and positive answers are scored as "1". On the positively worded items (4 to 6, social loneliness), the neutral and negative answers are scored as "1". Total score ranges from 0 (least lonely) to 6 (most lonely).

CONTACTS AND LOCATIONS:
Overall Officials: Tatia Mei-chun LEE, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No